CLINICAL TRIAL: NCT02902211
Title: Improving Mobility in Peripheral Artery Disease Using an Ankle Foot Orthosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0485-16-FB
Record Dates: First submitted 2016-08-24; First posted 2016-09-15 (Estimated); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Artery Disease
Keywords: ankle foot orthosis; biomechanics; mobility
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ankle foot orthosis (Experimental): Patients will wear an off-the-shelf, carbon composite AFO that is adjusted for them for three months. The patients will be asked to wear the AFO at all times except when they are in bed or showering/bathing. The instructions given to the patients about walking will be to follow the instructions from their doctor regarding risk factor management and exercise.
  Interventions: Device: Ankle foot orthosis
- Control (Active Comparator): Patients will be asked to follow the instructions from their doctor regarding risk factor management and exercise for three months.
  Interventions: Other: Control/standard of care

INTERVENTIONS:
Device: Ankle foot orthosis — Patients will wear an ankle foot orthosis at all times except when he/she is sleeping or bathing for three months.
  Arms: Ankle foot orthosis
Other: Control/standard of care — Patients will carry out with typical activities suggested by their physician for three months.
  Arms: Control

SUMMARY:
This study will determine whether an ankle foot orthosis (AFO) improves walking performance in participants with PAD from its first use. Additionally, the study will test walking performance after a three month AFO intervention and will examine the feasibility of this AFO intervention.

Data for evaluations will be collected from 50 participants with PAD. Fifty healthy age-matched controls will be participate in one baseline gait assessment for comparison purposes. Both groups between 40-85 years old.

Interventions and Evaluations Biomechanics evaluations: Patients with PAD will complete a biomechanics evaluation at baseline, following three months of control (standard of care), and following three months of AFO intervention. The evaluation will include measurement of walking distances, gait function, physical activity, quality of life, energy cost, muscle morphometrics, muscle activity, muscle oxygenation, and muscle strength and endurance while walking with and without the AFO. Healthy controls will be assessed during one baseline collection only and their participation in the study will then be finished.

Feasibility interview: All patients with PAD will participate in feasibility interviews that will assess acceptability, demand, implementation, and practicality. Interviews will occur 1.5 months and following completion of the AFO intervention (not the control arm).

AFO and Control (standard of care) Intervention: Patients will wear an off-the-shelf, carbon composite AFO that is adjusted to fit for three months. The patients will be asked to wear the AFO at all times except when they are in bed or showering/bathing. The instructions given to the patients about walking will be to follow the instructions from their doctor regarding risk factor management and exercise. The intervention order will be randomized and all subjects will participate in both arms.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a common cardiovascular disease manifesting from atherosclerotic blockages in the arteries of the legs. The most prevalent symptom of PAD is intermittent claudication, defined as pain or discomfort in the legs that is produced by physical activity and is relieved only through rest. PAD results in significant functional limitations such as slower walking velocity and an overall sedentary lifestyle. Prior research has documented significant deficits in gait biomechanics; specifically, an inability of the ankle plantar flexors to generate normal torque and power. Furthermore, insufficient blood flow was not found to be the only mechanism contributing to gait dysfunction in patients with PAD, but the affected muscle also demonstrates a myopathy that prevents normal leg function in these patients. Thus, treatment must consider muscular function and hemodynamics to improve function and increase activity levels. Supervised treadmill walking exercise is an effective treatment for increasing the distances patients with PAD can walk. However, there is a critical treatment gap for individuals whose disease presentations warrant a non--operative treatment plan but lack the motivation, time, access and monetary resources for supervised therapy. An ankle--foot orthosis (AFO) to offset ankle plantar flexor torque and power deficiency is a novel approach to increase the walking distances and physical activity levels in those with PAD. Made of a carbon-- composite material, AFOs are adjustable, affordable and could be prescribed and worn long--term to overcome the reduced propulsion and improve walking economy. The spring--like properties of carbon--composite AFOs allow energy storage at weight acceptance and return at the point of toe off, when the ankle plantar flexors are supposed to propel into the next step. Improvements in ankle kinetics and angular momentum have been reported by using an AFO with stroke, and other neuromuscular disorders affecting the legs. However, AFOs are typically worn for foot drop, and have never been implemented in patients with PAD to improve forward propulsion. Pilot work has shown that walking with an AFO instantly increases the initial and absolute walking distances in patients with PAD as much as pharmacotherapy for six months. An AFO addresses both the myopathy and low blood flow problems associated with claudication. Mechanical force from the AFO compensates for the insufficient propulsion force of the myopathic gastrocnemius muscles, while at the same time decreasing blood flow demand and muscular stress effects of ischemia. Thus an AFO allows patients to walk longer without pain or walk the distance needed to complete daily activities with less stress to the affected leg, and may preserve/improve the overall health of the PAD limb by lowering oxygen demands to PAD muscle and effort induced ischemia and stress.

Hypothesis: An AFO improves walking performance in patients with PAD by reducing the energy cost of walking and these improvements can be seen from the first time the patient uses the AFO. Further, an AFO intervention improves walking performance by improving the muscular function of patients' affected legs.

Specific Aim 1: Test the hypothesis that from its first use an AFO produces improvements in walking performance of patients with PAD by decreasing the required muscle contribution and energy cost of walking.

Specific Aim 2: Test the hypothesis that using an AFO for three months leads to progressive improvements in walking performance, physical activity levels and quality of life of patients with PAD and that these improvements correlate with improvements in the morphometric measurements, oxygenation levels, and muscle strength and endurance characteristics of the affected legs. A crossover design will be used, in which half of subjects will complete a three--month control period before, and half after, the AFO intervention.

Specific Aim 3: To determine the feasibility of a three month AFO intervention by examining acceptability (satisfaction, intent to continue use), demand (actual use, perceived demand), implementation (degree of use, success or failure of use, factors affecting use), and practicality (effects, ability of participants to use AFO).

If the hypothesis is correct, the study will be the first to demonstrate that a simple, accessible AFO device can rapidly improve functional status and quality of life in patients with PAD immediately by decreasing the required muscular contribution and oxygen demands to PAD muscle. Additionally, Aim #2 will evaluate the long--term effects of wearing an AFO on functional status and quality of life. Aim #3 will help the investigative team ensure it is feasible to implement the AFO in our target population. Detailed measures of mechanisms related with walking performance, muscle contribution, physical activity, quality of life and how these mechanisms change after wearing the AFO for three months will provide the evidence required to implement an AFO therapy that will improve functional status and quality of life in individuals with PAD.

ELIGIBILITY:
Inclusion Criteria:

* able to give written, informed consent
* demonstrate positive history of chronic claudication
* demonstrate exercise limiting claudication established by history and direct observation
* have an ankle/brachial index < 0.90 at rest
* have a stable blood pressure regimen, stable lipid regimen, stable diabetes regimen and risk factor control for 6 weeks.

Exclusion Criteria:

* rest pain or tissue loss due to PAD (Fontaine stage III and IV)2)
* acute lower extremity ischemic event secondary to thromboembolic disease or acute trauma
* walking capacity limited by conditions other than claudication including leg (joint/musculoskeletal, neurologic) and systemic (heart, lung disease) pathology

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Myers, PhD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Omaha VA Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan for our clinical trial involves making anonymized data sets available to qualified researchers to foster transparency, validate results, and facilitate secondary analyses. We will share raw and processed data, including baseline characteristics, outcome measures, adverse event reports, and accompanying metadata and documentation, such as data dictionaries and study protocols. Data will be available upon request through a formal application process to researchers affiliated with reputable institutions, contingent upon approval by an independent review committee and adherence to data use agreements to protect confidentiality and compliance with ethical standards.
Supporting Information: Study Protocol
Time Frame: Data will be available for five years upon the completion of the study.
Access Criteria: contact PI, samyers@unomaha.edu

REFERENCES:
- [Derived] Bashir AZ, Dinkel DM, Pipinos II, Estabrooks PA, Johanning JM, Myers SA. Long-term use of an ankle-foot orthosis intervention in patients with peripheral artery disease using the integrated promoting action on research implementation in health services (i-PARIHS) framework. Int J Cardiol. 2023 Feb 1;372:23-32. doi: 10.1016/j.ijcard.2022.11.041. Epub 2022 Nov 29. PMID 36455699

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were enrolled withdrew prior to randomization
Groups:
- Ankle Foot Orthosis Then Control: Patients will wear an off-the-shelf, carbon composite AFO that is adjusted for them for three months. The patients will be asked to wear the AFO at all times except when they are in bed or showering/bathing. The instructions given to the patients about walking will be to follow the instructions from their doctor regarding risk factor management and exercise.
  Ankle foot orthosis: Patients will wear an ankle foot orthosis at all times except when he/she is sleeping or bathing for three months.
- Control Then Ankle Foot Orthoses: Patients will be asked to follow the instructions from their doctor regarding risk factor management and exercise for three months.
  Control/standard of care: Patients will carry out with typical activities suggested by their physician for three months.
Period: First Three Months
Arm/Group | Ankle Foot Orthosis Then Control | Control Then Ankle Foot Orthoses
Started | 12 | 21
Completed | 5 | 18
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 7 | 3
Period: Second Three Months
Arm/Group | Ankle Foot Orthosis Then Control | Control Then Ankle Foot Orthoses
Started | 5 | 18
Completed | 2 | 13
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Control Then Ankle Foot Orthosis: Patients will be asked to follow the instructions from their doctor regarding risk factor management and exercise for three months.
  Control/standard of care: Patients will carry out with typical activities suggested by their physician for three months.
- Total: Total of all reporting groups
Arm/Group | Ankle Foot Orthosis Then Control | Control Then Ankle Foot Orthosis | Total
Number analyzed (Participants) | 12 | 21 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 8 | 18 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (6.2) | 72.6 (6.1) | 70.45 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 11 | 21 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 10 | 20 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 21 | 33
Claudication time (walking with AFO-Baseline) [Mean (Standard Deviation); unit: seconds]
  Initial claudication time (AFO) | 114.08 (71.91) | 190 (142.41) | 162.39 (125.81)
  Absoluteclaudication time (AFO) | 264.75 (227.03) | 322.3 (181.11) | 301.42 (197.5)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Walking Time From the Gardner Graded Treadmill Protocol
Description: Change in Initial claudication and the absolute claudication time from the progressive treadmill test when walking with ankle foot orthoses (AFO)
Time Frame: After three months of intervention with the ankle foot orthosis.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Ankle Foot Orthosis Then Control | Control Then Ankle Foot Orthosis
Number analyzed (Participants) | 4 | 14
Seconds
  Change in Initial walking time (First Intervention: 3 months) | 117.7 (89.8) | 197.5 (154.5)
  Change in Absolute walking time (Second Intervention: 3 months) | 188 (171.7) | 339.9 (171.5)

ADVERSE EVENTS:
Time Frame: Four weeks for each intervention.
Description: The number of participants at risk for Other (Not Including Serious) Adverse Events is thirty-three; however, throughout the course of the trial, none of them experienced any instances of such adverse events reported among the participants. This indicates that none of the participants experienced any adverse events.
Arm/Group | Ankle Foot Orthosis | Control
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT02902211/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT02902211/ICF_001.pdf